CLINICAL TRIAL: NCT07221071
Title: Supporting Women With Breast Cancer to Prepare for Treatment (The Prepare Study)
Acronym: Prepare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Katharine Yao, MD, Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EH20-134
Record Dates: First submitted 2025-10-21; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Mindfulness
Keywords: Cancer Surgery; Mindfulness; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Arm (Experimental): Brief video and audio practice of mindfulness
  Interventions: Behavioral: Mindfulness Arm
- Health Videos - Mike Evans (Placebo Comparator): Brief videos focusing on health and wellness
  Interventions: Other: Control group placebo

INTERVENTIONS:
Behavioral: Mindfulness Arm — Participants will be instructed to watch four brief breast cancer specific educational mindfulness videos (within the first week of randomization), listen to guided audio recordings of different mindfulness meditations at least 3 times per week throughout the intervention period (which lasts until the Time 3 Assessment), and complete brief, post-listening written reflections in a journal (NOW reflections) that is provided to them during the intervention period.
  Arms: Mindfulness Arm
Other: Control group placebo — Participants will receive brief videos that focuses on general health behaviors. We will utilize the Mike Evans chalkboard videos (https://www.reframehealthlab.com/category/whiteboard-health-videos/) as the control for this group. Participants will view the Mike Evans videos within the first week following randomization. The participants will be assigned to watch 10 videos located on the Group B study website. Topics range from cancer fatigue, healthy eating, benefits of exercise, and the science of happiness.
  Arms: Health Videos - Mike Evans

SUMMARY:
The purpose of this study is to evaluate if a brief mindfulness intervention before and after surgery would impact patient emotional wellbeing, quality of life, and biomarkers measured before and after surgery by finger prick collection and surveys.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate a brief, technology-enabled mindfulness intervention before and following breast cancer surgery to determine its impact on emotional wellbeing and biological stress response in breast cancer patients. The investigators will administer self-reported questionnaires of emotional wellbeing and quality of life and collect pro and anti-inflammatory cytokines (CRP and IL-10, respectively) using a minimally invasive finger prick approach. The findings from this study will help establish an evidence base on the efficacy of a brief, technology enabled mindfulness intervention on patient anxiety, wellbeing and biological response. No previous studies have examined the impact of a brief mindfulness training prior to and following surgery on patient wellbeing. The long-term goal is to determine whether brief, technology-enabled mindfulness support can become part of routine preparation for breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Females >20 and < 85 years of age
2. History of contralateral breast cancer in the past is acceptable
3. Patients seeking second opinion for diagnosis are eligible
4. Clinical AJCC stage 0-III breast cancer
5. Patients who have an in breast tumor recurrence are eligible
6. English Speaking
7. Willing to fill out surveys required for the study
8. Gene mutation carriers are eligible
9. Neoadjuvant therapy patients are eligible

Exclusion Criteria:

1. AJCC Stage IV breast cancer
2. Unwilling to fill out surveys for the study
3. Patients with a distant recurrence
4. Patients unaware of their diagnosis

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Anxiety | 3 months
  To measure the impact of a mindfulness intervention instituted prior to surgery on patient anxiety for newly diagnosed breast cancer patients, using the PROMIS anxiety questionnaire [Emotional Distress - Anxiety - Short Form 8a answer options are: Never, Rarely, Sometimes, Often, Always].

SECONDARY OUTCOMES:
Patient Depression | 3 months
  To measure the impact of a mindfulness intervention on patient depression using the [PROMIS Emotional Distress - Depression - Short Form 8a questionnaire - options are Never, Rarely, Sometimes, Often, Always].
Psychosocial wellbeing | 3 months
  To compare psychosocial wellbeing as it pertains to body image between those receiving a mindfulness intervention or general overall health videos, by using the Breast Q questionnaire - answer options are: None of the time, A little of the time, some of the time, most of the time, and all of the time.
Stress biomarker | 3 months
  To determine if a mindfulness intervention will impact stress biomarker profiles. Participants will be asked to provide self-collected whole dried blood spots to assess IL-6, CRP, and TNF-α using a minimally invasive finger skin prick technique, which involves pricking the finger with a lancet, milking the finger to produce 5 drops of blood onto filter paper, allowing the blood spots to dry, and mailing it to the study team at MGH in a secure envelope.

OTHER OUTCOMES:
Exploratory | 3 months
  To determine if a mindfulness intervention will impact patient fear of recurrence, using a fear of recurrence questionnaire - answer options are strongly disagree, disagree, not certain, agree, strongly agree.
Self-Kindness questionnaire | 3 months
  To measure patient self- compassion and kindness. using a (Self-Compassion Scale-5 items- answer choices are: Almost Never, Never, Sometimes, Always, Almost Always)
Emotional Reactivity/Regulation and Mindfulness Awareness | 3 months
  Patients will complete the Nonreactivity scale (Five Facet Mindfulness Questionnaire-7 items - answer choices are: Never or very rarely true, Rarely true, Sometimes true, Often true, and Very often true or always true).

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Yao, M.D, Principal Investigator — Endeavor Health
Locations (1):
- Endeavor Health, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black DS, Slavich GM. Mindfulness meditation and the immune system: a systematic review of randomized controlled trials. Ann N Y Acad Sci. 2016 Jun;1373(1):13-24. doi: 10.1111/nyas.12998. Epub 2016 Jan 21. PMID 26799456
- [Background] Bishop SR, Lau M, Shapiro S, et al. Mindfulness: A Proposed Ooperational Definition. Clinical Psychology: Science and Practice. 2004;11(3):230-241